CLINICAL TRIAL: NCT00990821
Title: A Randomized, 5-Part, Intravenous Study of the Safety, Tolerability, Bioequivalence, and Drug Interaction Potential of Final Market Image Formulation of MK0517 in Young Healthy Subjects
Brief Title: A Study to Investigate the Safety and Tolerability of MK-0517 in Healthy Subjects (MK-0517-012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0517-012; MK-0517-012
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Results first posted 2013-12-12 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Vomiting; Postoperative Nausea and Vomiting | interventions — Aprepitant; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (14):
- Part I, Panel A (Experimental): 100 mg MK-0517 (nonpolysorbate 80 formulation [non-PS80]) or placebo → 150 mg MK-0517 (non- PS80) or placebo → 125 mg aprepitant
  Interventions: Drug: 100 MK-0517 (PS80) + 2 mg midazolam; Drug: 100 mg MK-0517 (non-PS80); Drug: 150 mg MK-0517 (Non-PS80); Drug: Placebo; Drug: 125 mg Aprepitant
- Part I, Panel B (Experimental): 100 mg MK-0517 (PS80 formulation [PS80]) or placebo → 150 mg MK-0517 (PS80) or placebo → 125 mg aprepitant
  Interventions: Drug: 100 mg MK-0517 (PS80); Drug: 150 mg MK-0517 (PS80); Drug: Placebo; Drug: 125 mg Aprepitant
- Part I, Panel C (Experimental): 40 mg MK-0517 (non-PS80) or placebo → 40 mg aprepitant
  Interventions: Drug: 40 mg MK-0517 (non-PS80); Drug: Placebo; Drug: 40 mg Aprepitant
- Part II (Experimental): 2 mg midazolam → 100 mg MK-0517 (PS80) + 2 mg midazolam
  Interventions: Drug: 100 mg MK-0517 (PS80); Drug: 2 mg Midazolam
- Part III, Panel 1, Treatment Sequence 1 (Experimental): 125 mg aprepitant → 90 mg MK-0517 (PS80)
  Interventions: Drug: 90 mg MK-0517 (PS80); Drug: 40 mg MK-0517 (non-PS80); Drug: 125 mg Aprepitant
- Part III, Panel 1, Treatment Sequence 2 (Experimental): 40 mg MK-0517 (non-PS80) → 125 mg aprepitant
  Interventions: Drug: 40 mg MK-0517 (non-PS80); Drug: 125 mg Aprepitant
- Part III, Panel 2 (Experimental): 40 mg MK-0517 (non-PS80)
  Interventions: Drug: 40 mg MK-0517 (non-PS80)
- Part IV (Experimental): 40 mg MK-0517 (non-PS80 formulation)
  Interventions: Drug: 40 mg MK-0517 (non-PS80)
- Part V, Treatment Sequence 1 (Experimental): 125 mg aprepitant → 100 mg MK-0517 (PS80) → 115 mg MK-0517 (PS80 formulation)
  Interventions: Drug: 100 mg MK-0517 (PS80); Drug: 115 mg MK-0517 (PS80); Drug: 125 mg Aprepitant
- Part V, Treatment Sequence 2 (Experimental): 100 mg MK-0517 (PS80) → 115 mg MK-0517 (PS80) → 125 mg aprepitant
  Interventions: Drug: 100 mg MK-0517 (PS80); Drug: 115 mg MK-0517 (PS80); Drug: 125 mg Aprepitant
- Part V, Treatment Sequence 3 (Experimental): 115 mg MK-0517 (PS80) → 125 mg aprepitant → 100 mg MK-0517 (PS80)
  Interventions: Drug: 100 mg MK-0517 (PS80); Drug: 115 mg MK-0517 (PS80); Drug: 125 mg Aprepitant
- Part V, Treatment Sequence 4 (Experimental): 125 mg aprepitant → 115 mg MK-0517 (PS80) → 100 mg MK-0517 (PS80)
  Interventions: Drug: 100 mg MK-0517 (PS80); Drug: 115 mg MK-0517 (PS80); Drug: 125 mg Aprepitant
- Part V, Treatment Sequence 5 (Experimental): 100 mg MK-0517 (PS80) → 125 mg aprepitant → 115 mg MK-0517 (PS80)
  Interventions: Drug: 100 mg MK-0517 (PS80); Drug: 115 mg MK-0517 (PS80); Drug: 125 mg Aprepitant
- Part V, Treatment Sequence 6 (Experimental): 115 mg MK-0517 (PS80) → 100 mg MK-0517 (PS80) → 125 mg aprepitant
  Interventions: Drug: 100 mg MK-0517 (PS80); Drug: 115 mg MK-0517 (PS80); Drug: 125 mg Aprepitant

INTERVENTIONS:
Drug: 90 mg MK-0517 (PS80) — MK-0517 (PS80 formulation), 1 mg/mL, administered intravenous (IV) over 15 minutes
  Arms: Part III, Panel 1, Treatment Sequence 1
Drug: 100 mg MK-0517 (PS80) — MK-0517 (PS80 formulation), 1 mg/mL, administered IV over 15 minutes
  Arms: Part I, Panel B; Part II; Part V, Treatment Sequence 1; Part V, Treatment Sequence 2; Part V, Treatment Sequence 3; Part V, Treatment Sequence 4; Part V, Treatment Sequence 5; Part V, Treatment Sequence 6
Drug: 100 MK-0517 (PS80) + 2 mg midazolam — MK-0517 (Non-PS80 formulation), 1 mg/mL, administered IV over 15 minutes. Midazolam is co-administered as a single oral 2-mg dose of midazolam with MK-0517.
  Arms: Part I, Panel A
Drug: 115 mg MK-0517 (PS80) — MK-0517 (PS80 formulation), 1 mg/mL, administered IV over 15 minutes
  Arms: Part V, Treatment Sequence 1; Part V, Treatment Sequence 2; Part V, Treatment Sequence 3; Part V, Treatment Sequence 4; Part V, Treatment Sequence 5; Part V, Treatment Sequence 6
Drug: 150 mg MK-0517 (PS80) — MK-0517 (PS80 formulation), 1 mg/mL, administered IV over 15 minutes
  Arms: Part I, Panel B
Drug: 40 mg MK-0517 (non-PS80) — MK-0517 (Non-PS80) is administered as single IV dose over 30 seconds.
  Arms: Part I, Panel C; Part III, Panel 1, Treatment Sequence 1; Part III, Panel 1, Treatment Sequence 2; Part III, Panel 2; Part IV
Drug: 100 mg MK-0517 (non-PS80) — MK-0517 (Non-PS80) is administered as single IV dose over 30 seconds.
  Arms: Part I, Panel A
Drug: 150 mg MK-0517 (Non-PS80) — MK-0517 (Non-PS80) is administered as single IV dose over 30 seconds.
  Arms: Part I, Panel A
Drug: Placebo — Placebo matching MK-0517
  Arms: Part I, Panel A; Part I, Panel B; Part I, Panel C
Drug: 40 mg Aprepitant — Aprepitant, oral, tablet, single dose
  Arms: Part I, Panel C
Drug: 125 mg Aprepitant — Aprepitant oral tablet, single dose
  Arms: Part I, Panel A; Part I, Panel B; Part III, Panel 1, Treatment Sequence 1; Part III, Panel 1, Treatment Sequence 2; Part V, Treatment Sequence 1; Part V, Treatment Sequence 2; Part V, Treatment Sequence 3; Part V, Treatment Sequence 4; Part V, Treatment Sequence 5; Part V, Treatment Sequence 6
Drug: 2 mg Midazolam — Midazolam oral tablet, single dose
  Arms: Part II

SUMMARY:
This 5-part study will evaluate the safety, tolerability, and pharmacokinetics of two formulations of MK-0517 (with and without polysorbate 80) and aprepitant in healthy adults. Parts I to IV of this study will examine different doses of MK-0517 as well as two different formulations of MK-0517 (with and without polysorbate 80). Part V of the study will compare single doses of intravenous non-PS80 MK-0517 to oral 125-mg capsule of aprepitant. The primary hypothesis for Part V of the study is that a single intravenous dose of 100-mg or 115-mg MK-0517 is area under the plasma-time curve (AUC) equivalent to that of the 125-mg oral aprepitant capsule in young healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Subject is neither grossly overweight nor underweight for his/her height and body build
* Subject is in good health -Subject is a nonsmoker
* Subject is willing to avoid excessive alcohol consumption for the duration of the study
* Subject is willing to avoid strenuous physical activity (i.e. unaccustomed weight lifting, running, bicycling) for the duration of the study
* Subject agrees to refrain from consumption of grapefruit (and grapefruit products) before and during the study

Exclusion Criteria:

* Subject has a history of multiple and/or severe allergies to drugs or food
* Subject has donated blood or taken an investigational drug in another clinical trial within the last 4 weeks
* Subject has an infection, including Human immunodeficiency virus (HIV) infection
* Subject is a regular user of any illicit drug
* Subject consumes excessive amounts of alcohol
* Subject drinks excessive amounts of coffee, tea, cola or other caffeinated beverages
* Subject currently uses on a regular basis, any prescription or non prescription medications

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One Investigator in the United States. Primary therapy period: 31-Jan-2005 to 01-Dec-2005.
Groups:
- Part I, Panel A: 100 mg MK-0517 (non-polysorbate 80 formulation [non-PS80]) or placebo → 150 mg MK-0517 (non-PS80) or placebo → 125 mg aprepitant
Period: Overall Study
Arm/Group | Part I, Panel A | Part I, Panel B | Part I, Panel C | Part II | Part III, Panel 1, Treatment Sequence 1 | Part III, Panel 1, Treatment Sequence 2 | Part III, Panel 2 | Part IV | Part V, Treatment Sequence 1 | Part V, Treatment Sequence 2 | Part V, Treatment Sequence 3 | Part V, Treatment Sequence 4 | Part V, Treatment Sequence 5 | Part V, Treatment Sequence 6
Started | 14 | 16 | 14 | 8 | 17 | 17 | 12 | 14 | 12 | 14 | 12 | 14 | 12 | 12
Completed | 14 | 14 | 14 | 8 | 14 | 14 | 11 | 14 | 12 | 13 | 9 | 9 | 10 | 11
Not Completed | 0 | 2 | 0 | 0 | 3 | 3 | 1 | 0 | 0 | 1 | 3 | 5 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 3 | 3 | 1 | 0 | 0 | 1 | 3 | 5 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I, Panel A | Part I, Panel B | Part I, Panel C | Part II | Part III, Panel 1, Treatment Sequence 1 | Part III, Panel 1, Treatment Sequence 2 | Part III, Panel 2 | Part IV | Part V, Treatment Sequence 1 | Part V, Treatment Sequence 2 | Part V, Treatment Sequence 3 | Part V, Treatment Sequence 4 | Part V, Treatment Sequence 5 | Part V, Treatment Sequence 6 | Total
Number analyzed (Participants) | 14 | 16 | 14 | 8 | 17 | 17 | 12 | 14 | 12 | 14 | 12 | 14 | 12 | 12 | 188
Age, Continuous [Mean (Full Range); unit: years] | 31.2 [21 to 45] | 35.2 [23 to 44] | 33.1 [22 to 45] | 36.9 [25 to 45] | 33.2 [19 to 43] | 33.2 [19 to 43] | 32.4 [18 to 45] | 29.4 [18 to 45] | 31.9 [19 to 44] | 33.5 [22 to 44] | 31.3 [22 to 45] | 29.1 [19 to 41] | 30.4 [19 to 45] | 36.5 [20 to 43] | 32.6 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 10 | 5 | 11 | 10 | 10 | 10 | 7 | 11 | 6 | 6 | 4 | 6 | 112
  Male | 7 | 7 | 4 | 3 | 6 | 7 | 2 | 4 | 5 | 3 | 6 | 8 | 8 | 6 | 76

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma-Time Curve (AUC[0 to Infinity]) for Aprepitant and MK-0517 for Study Part V
Description: AUC (0-inf) is the area under the plasma concentration-time curve from time zero extrapolated to infinite time. The AUC(0-inf) bioequivalence was evaluated for single doses of 100 and 115 mg MK-0517 PS80, IV and that of an oral 125-mg capsule of aprepitant. Period I to IV populations are not included in the outcome analysis because those were formulation and dose-finding/dose confirmation arms.
Time Frame: Up to 72 Hours Post Dose
Population: All participants in Part V who had at least one period of AUC data were included in the evaluation of pharmacokinetics. Participants without sufficient concentration data for an AUC calculation included: 6 participants in the Aprepitant (125 mg) , 8 participants in the MK-0517 (100 mg) group, and 5 participants in the MK-0517 (115 mg) group.
Measure: Least Squares Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Aprepitant (125 mg): A single oral dose with an Aprepitant capsule
- MK-0517 (100 mg): 100 mg of MK0517 (PS80 formulation) as an IV (intravenous) administered over 15 minutes
- MK-0517 (115 mg): 115 mg of MK0517 (PS80 formulation) as an IV (intravenous) administered over 15 minutes
Arm/Group | Aprepitant (125 mg) | MK-0517 (100 mg) | MK-0517 (115 mg)
Number analyzed (Participants) | 70 | 68 | 71
ng*hr/mL | 29215 (15731) | 24961 (10477) | 31724 (14287)

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study drug
Description: All 188 study participants are included in the safety population: Adverse events are reported for the actual doses given in any part of the study. Individual participants may have received more than one drug or more than one dose of a drug.
Groups:
- 90 mg MK-0517 (PS80); 100 mg MK-0517 (PS80); 115 mg MK-0517 (PS80); 150 mg MK-0517 (PS80); 100 mg MK-0517 (Non-PS80); 150 mg MK-0517 (Non-PS80): MK-0517, PS80 formulation, administered with a single IV administration
- 100 mg MK-0517 (PS80) + 2 mg Midazolam: PS80 formulation, administered with a single IV administration and a single oral administration of midazolam
- 40 mg MK-0517 (Non-PS80): MK-0517, non-PS80 formulation, administered with a single IV administration
- Placebo: Placebo matching MK-0517 (PS80 or non-PS80)
- 40 mg Aprepitant: Aprepitant administered by a single oral capsule
- 125 mg Aprepitant: Aprepitant administered as a single oral capsule
- 2 mg Midazolam: Midazolam administered as a single oral solution
Arm/Group | 90 mg MK-0517 (PS80) | 100 mg MK-0517 (PS80) | 100 mg MK-0517 (PS80) + 2 mg Midazolam | 115 mg MK-0517 (PS80) | 150 mg MK-0517 (PS80) | 40 mg MK-0517 (Non-PS80) | 100 mg MK-0517 (Non-PS80) | 150 mg MK-0517 (Non-PS80) | Placebo | 40 mg Aprepitant | 125 mg Aprepitant | 2 mg Midazolam
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/82 | 0/8 | 0/66 | 0/12 | 0/36 | 0/12 | 0/11 | 0/11 | 0/14 | 0/133 | 0/8
Other Adverse Events (participants affected / at risk) | 8/31 | 8/82 | 5/8 | 7/66 | 3/12 | 4/36 | 3/12 | 6/11 | 2/11 | 2/14 | 6/133 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 90 mg MK-0517 (PS80) (N=31) | 100 mg MK-0517 (PS80) (N=82) | 100 mg MK-0517 (PS80) + 2 mg Midazolam (N=8) | 115 mg MK-0517 (PS80) (N=66) | 150 mg MK-0517 (PS80) (N=12) | 40 mg MK-0517 (Non-PS80) (N=36) | 100 mg MK-0517 (Non-PS80) (N=12) | 150 mg MK-0517 (Non-PS80) (N=11) | Placebo (N=11) | 40 mg Aprepitant (N=14) | 125 mg Aprepitant (N=133) | 2 mg Midazolam (N=8)
Induration (General disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 1 | 4 | 0 | 1 | 2 | 2 | 5 | 0 | 0 | 0 | 0
Infusion Site Pain (General disorders) | 0 | 7 | 1 | 5 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 0 | 0 | 2 | 2 | 0 | 0 | 3 | 2 | 0 | 5 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intraocular Pressure Test (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eye Irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.